CLINICAL TRIAL: NCT05083988
Title: Effect of Virtual Reality Distraction Versus Audio Distraction on Anxiety and Pain Reduction in Children Undergoing Dental Treatment (A Randomized Clinical Trial)
Brief Title: Effect of Virtual Reality Distraction on Anxiety and Pain Reduction in Children Undergoing Dental Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omneya Ahmed AbdelRazik saleh, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Dental anxiety reduction
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: parallel-group and allocation ratio (1:1) Intervention: virtual reality glasses. Control: audiodistraction using music
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- audiovisual distraction (Experimental)
  Interventions: Device: virtual reality glasses
- audiodistraction (Experimental)
  Interventions: Device: music

INTERVENTIONS:
Device: virtual reality glasses — a system composed of a head-mounted wide view display placed in front of the eyes and headphones placed in ears, it has the ability to block the real-world stimuli. This could distract the patient from the dental environment, which helps reduce anxiety
  Other Names: audiovisual distraction
  Arms: audiovisual distraction
Device: music — Music can be used to distract patients from the anxiety provoking stimulus. It helps the patient to escape from the stressful reality as it activates imaginary. Psychosocially music can offer peace and comfort to patients during dental treatment as it helps in making the environment less threatening.
  Other Names: audiodistraction
  Arms: audiodistraction

SUMMARY:
The aim of the study is to evaluate and compare the effect of virtual reality glasses (VR) as an audiovisual distraction method to audio distraction using music on child's dental anxiety during dental treatment.

DETAILED DESCRIPTION:
a randomized clinical trial with parallel-group and allocation ratio (1:1). intervention group: audiovisual distraction using virtual reality glasses control group :audio distraction using music. in children aged 5-8 years who need dental extraction for primary molars.

For both groups:

1. Taking personal data, medical and dental history.
2. Diagnosis and determination of the required treatment.
3. Measuring preoperative anxiety (expressed by heart rate) using a pulse oximeter.
4. Using the behavior guidance technique:

   Intervention group: The Child is introduced to the virtual reality glasses device, and was given instructions on how to use it and was allowed to choose one of previously chosen cartoons to be played during the procedure.

   Control group: The child is introduced to the headphones and was given instructions on how to use it, and a relaxing music is played during the procedure.
5. Administration of topical anesthesia.
6. Administration of local anesthesia.
7. Check the effectiveness of local anesthesia using dental probe.
8. Extraction of the affected tooth.
9. Measuring postoperative anxiety (expressed by heart rate) using the pulse oximeter.
10. Evaluate the objective pain using Face, Legs, Cry, Consolabiliy scale .
11. Self-reporting of subjective pain using Visual analogue scale.
12. Post extraction instructions are given to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-8 years.
* Children without any mental or systemic disorder.
* Children need extraction of primary molars under local anesthesia.

Exclusion Criteria:

* Children with visual impairment.
* Children with hearing disabilities.
* Patients or caregivers who refuse to sign the consent.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
preoperative anxiety | before administration of local anesthesia
  Preoperative anxiety will be measured before administration of local anesthesia using a fingertip pulse oximeter in beat per minute unit (BPM)
postoperative anxiety | immediately after dental extraction
  using a fingertip pulse oximeter in beat per minute unit (BPM)
preoperative anxiety | before administration of local anesthesia
  RMS-pectorial scale ( Raghavendra, Madhuri, Sujata - pectorial scale) before administration of local anesthesia in a numerical unit from 1-5 where 1 denotes the minimum anxiety and 5 denotes the maximum anxiety
postoperative anxiety | immediately after dental extraction
  S-pectorial scale ( Raghavendra, Madhuri, Sujata - pectorial scale) immediatly after extraction in a numerical unit from 1-5 where 1 denotes the minimum anxiety and 5 denotes the maximum anxiety

SECONDARY OUTCOMES:
subjective pain | immediately after extraction.
  using Visual analogue scale (vas scale) (0-10) , self reported pain as the child choose a number from 0 to 10 which describes the intensity of his or her pain.
  0 =no pain 10=extreme pain.
objective pain | during dental extraction procedure.
  using FLCCS (0-10)valuated by the outcomes assessor. The FLACC scale has five criteria - Faces, Legs, Activity, Cry, Consolability, which are each assigned a score of 0, 1 or 2. Total score of scale is summed in range 0 to 10, where: 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] CustOdio NB, Cademartori MG, Azevedo MS, Mendes MA, Schardozim LR, Costa LRRSD, Goettems ML. Efficacy of audiovisual distraction using eyeglasses during dental care: a randomized clinical trial. Braz Oral Res. 2021 Feb 12;35:e26. doi: 10.1590/1807-3107bor-2021.vol35.0026. eCollection 2021. PMID 33605356
- [Result] Packyanathan JS, Lakshmanan R, Jayashri P. Effect of music therapy on anxiety levels on patient undergoing dental extractions. J Family Med Prim Care. 2019 Dec 10;8(12):3854-3860. doi: 10.4103/jfmpc.jfmpc_789_19. eCollection 2019 Dec. PMID 31879625
- [Result] Felemban OM, Alshamrani RM, Aljeddawi DH, Bagher SM. Effect of virtual reality distraction on pain and anxiety during infiltration anesthesia in pediatric patients: a randomized clinical trial. BMC Oral Health. 2021 Jun 25;21(1):321. doi: 10.1186/s12903-021-01678-x. PMID 34172032
- [Result] Nunna M, Dasaraju RK, Kamatham R, Mallineni SK, Nuvvula S. Comparative evaluation of virtual reality distraction and counter-stimulation on dental anxiety and pain perception in children. J Dent Anesth Pain Med. 2019 Oct;19(5):277-288. doi: 10.17245/jdapm.2019.19.5.277. Epub 2019 Oct 30. PMID 31723668
- [Result] Scheerman JFM, van Meijel B, van Empelen P, Kramer GJC, Verrips GHW, Pakpour AH, Van den Braak MCT, van Loveren C. Study protocol of a randomized controlled trial to test the effect of a smartphone application on oral-health behavior and oral hygiene in adolescents with fixed orthodontic appliances. BMC Oral Health. 2018 Feb 7;18(1):19. doi: 10.1186/s12903-018-0475-9. PMID 29415697
- [Result] Grisolia BM, Dos Santos APP, Dhyppolito IM, Buchanan H, Hill K, Oliveira BH. Prevalence of dental anxiety in children and adolescents globally: A systematic review with meta-analyses. Int J Paediatr Dent. 2021 Mar;31(2):168-183. doi: 10.1111/ipd.12712. Epub 2020 Sep 9. PMID 33245591
- [Result] Dahlander A, Soares F, Grindefjord M, Dahllof G. Factors Associated with Dental Fear and Anxiety in Children Aged 7 to 9 Years. Dent J (Basel). 2019 Jul 1;7(3):68. doi: 10.3390/dj7030068. PMID 31266156
- [Result] Raja SN, Carr DB, Cohen M, Finnerup NB, Flor H, Gibson S, Keefe FJ, Mogil JS, Ringkamp M, Sluka KA, Song XJ, Stevens B, Sullivan MD, Tutelman PR, Ushida T, Vader K. The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. Pain. 2020 Sep 1;161(9):1976-1982. doi: 10.1097/j.pain.0000000000001939. PMID 32694387
- [Result] Lopez-Valverde N, Muriel Fernandez J, Lopez-Valverde A, Valero Juan LF, Ramirez JM, Flores Fraile J, Herrero Payo J, Blanco Antona LA, Macedo de Sousa B, Bravo M. Use of Virtual Reality for the Management of Anxiety and Pain in Dental Treatments: Systematic Review and Meta-Analysis. J Clin Med. 2020 Apr 5;9(4):1025. doi: 10.3390/jcm9041025. PMID 32260538 (Retraction: PMID 32731319 J Clin Med. 2020 Jul 28;9(8):)
- [Result] Sivakumar P, Gurunathan D. Behavior of Children toward Various Dental Procedures. Int J Clin Pediatr Dent. 2019 Sep-Oct;12(5):379-384. doi: 10.5005/jp-journals-10005-1670. PMID 32440041